CLINICAL TRIAL: NCT01123109
Title: 3-D Endoanal Ultrasound: Normative Anatomy of the Anal Sphincter in Nulliparous Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Karen Noblett, Division Director, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2007-5983
Record Dates: First submitted 2010-05-06; First posted 2010-05-14 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Normal (no Known Injury) Anal Sphincter Female Anatomy
Keywords: nulliparous women

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nulliparous females (Other): nulliparous women over the age of 18
  Interventions: Procedure: 3-D Endoanal Ultrasound

INTERVENTIONS:
Procedure: 3-D Endoanal Ultrasound — The subject will be placed in the supine position with their feet in the stirrups and a drape will be used, exposing only the anus and perineum in order to introduce the probe. In order to prevent and minimize any potential discomfort, the lubricated ultrasound probe will be gently inserted into the anal canal up to the anal verge, with minimal manipulation of the probe once inserted. The scan lasts approximately two minutes and the entire exam will take no more than five minutes.

SUMMARY:
The purpose of this research study is to measure the muscles that make up your anal sphincter (muscles that control bowel movements) by using ultrasound. The most common way for women to injure these muscles is through childbirth. Some physicians think about 30% of women delivering their first baby develop some anal sphincter damage, which may or may not lead to symptoms such as anal urgency or incontinence (involuntary loss of gas or stool). The purpose of the study is to measure muscles in normal women who have never given birth or had an injury to their anal sphincter.

DETAILED DESCRIPTION:
Participants will be asked to complete a one page questionnaire. This questionnaire will address whether perineal trauma, sphincter lacerations, anal incontinence, and fecal urgency impact the subject on any level. Subjects will also be asked about their bowel habits and history of problems with bowel movements. Subjects will then be asked to undergo an ultrasound study of the anal sphincter at the time of enrollment. Completing the entire study will take no more than 15 minutes. This will be done at the doctor's office. Answering the questionnaire will take no more than 5 minutes.

The endoanal ultrasound is a probe with a diameter equivalent to the index finger. It is inserted in the rectum and measures the length and width of the sphincter muscles.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous women over the age of 18.

Exclusion Criteria:

* any history of anal incontinence, chronic constipation, anorectal disease or trauma, neuromuscular or neuropsychiatric disease, diabetes, gastrointestinal disorders, or previous anorectal or pelvic surgeries.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To establish normative data for the anal sphincter complex in asymptomatic nulliparous females without sphincter disruption sphincter. | 15 minute exam

CONTACTS AND LOCATIONS:
Overall Officials: Karen Noblett, MD, Principal Investigator — UCI Medical Center
Locations (1):
- UCI Women's Healthcare, Orange, California, United States